CLINICAL TRIAL: NCT07358741
Title: Balancing Time and Outcomes: A Prospective Observational Study Comparing the Effectiveness of the Standard Two-Day Advanced Life Support (ALS) Versus One Day Recertification Course
Brief Title: Standard Two-Day Advanced Life Support (ALS) Versus One Day Recertification Course
Status: Recruiting | Type: Observational
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, Associate professor-intensive care medicine, National Hepatology & Tropical Medicine Research Institute
Other Study IDs: NHTMRI-IRB-30-2025
Record Dates: First submitted 2025-12-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Skill Performance; Knowledge
Keywords: Standard; recertification; ALS; ERC; knowledge retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard ALS course: Two day course
- Recertification Course: one day course

SUMMARY:
this study aims to compare the effectiveness of a one-day versus two-day ALS recertification course in terms of knowledge retention, practical skills performance, participant satisfaction, and confidence.

DETAILED DESCRIPTION:
demographic data will be collected, including participants' age, sex, specialty, prior ALS course completion, participation in resuscitation teams, last CPR performance, and total online learning hours (minimum 16 hours for the standard ALS course and 8 hours for the recertification course). All ALS courses (standard and recertification) will be conducted in accordance with the standardized curriculum, structure, and educational formats established by the European Resuscitation Council (ERC).

Assessments:

A. Knowledge Assessment B. Practical Skills Performance C. Participant satisfaction and confidence at the end of each course

• Scoring: 0 = Not performed/incorrect, 1 = Partially/performed with prompting, 2 = Performed correctly and independently.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthcare professionals (≥18 years) requiring ALS recertification, including doctors, nurses, and paramedics, who can attend the assigned course and follow-up assessments.

Exclusion Criteria:

* Participants will be excluded if they cannot attend the assigned course or decline consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: demographic data will be collected, including participants' age, sex, specialty, prior ALS course completion, participation in resuscitation teams, last CPR performance, and total online learning hours (minimum 16 hours for the standard ALS course and 8 hours for the recertification course).
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
overall effectiveness between the two-day stanrdand one-day ALS recertification | 24hours precourse
  • Baseline knowledge score
Practical skill effectiveness | 48 and 24 hours from standard amd recertification course respectively
  • Standardized team-leader assessment station at the end of each course. Scoring: 0 = Not performed/incorrect, 1 = Partially/performed with prompting, 2 = Performed correctly and independently.
Knowledge retention assessment | 3 months post course
  post-course MCQ to evaluate decay; similar to pre-course MCQ

SECONDARY OUTCOMES:
Participant satisfaction e | 48hours and 24 from standard and recertification course respectively
  scores about course structure, teaching quality, and learning materials; 1: Strongly disagree- 2:disagree- 3: moderate 4: agree- 5: Strongly agree

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian resuscitation council, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) generated in this study will not be made publicly available in order to protect participant confidentiality and comply with ethical regulations.